CLINICAL TRIAL: NCT02111018
Title: Extracorporeal Therapy for the Removal of Myoglobin Using the CytoSorb in Patients With Rhabdomyolysis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: CytoSorbents, Inc (Industry)
Collaborators: San Antonio Military Medical Center (SAMMC), US Army Institute of Surgical Research-Burn Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CytoSorb 2013-001
Record Dates: First submitted 2014-03-19; First posted 2014-04-10 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVVH (Active Comparator)
  Interventions: Procedure: CVVH
- CytoSorb Device (Experimental)
  Interventions: Device: CytoSorb Device

INTERVENTIONS:
Device: CytoSorb Device
  Arms: CytoSorb Device
Procedure: CVVH
  Arms: CVVH

SUMMARY:
Prospective, randomized non-blinded, controlled study to assess the feasibility of the CytoSorb as an adjunct to the standard of care in patients with rhabdomyolysis requiring renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18-80
* Subjects present with rhabdomyolysis
* Subject requires renal replacement therapy and has undergone adequate volume resuscitation
* Subject is willing to comply with specified follow up requirements

Exclusion Criteria:

* Subject or their legal guardian either declines or cannot give informed consent
* Subject is pregnant
* Subject has been previously enrolled in this clinical study
* Comorbid condition that may limit survival to ≤14 days
* Comorbid condition that could confound study results
* Subjects who are receiving immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of device as measured by change in myoglobin | 30 days
Assessment of serious device or procedure-related adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: LTC Kevin Chung, MD, Principal Investigator — San Antonio Military Medical Center-US Army Institute of Surgical Research-Burn Center; MAJ Ian Stewart, MD, Principal Investigator — San Antonio Military Medical Center-US Army Institute of Surgical Research- Burn Center
Locations (1):
- San Antonio Military Medical Center- US Army Institute of Surgical Research- Burn Center, San Antonio, Texas, United States